CLINICAL TRIAL: NCT02573870
Title: 201546, A Repeat-dose Study of Batefenterol/FF (GSK961081/GW685698) Compared With Placebo in the Treatment of COPD
Brief Title: Batefenterol/Fluticasone Furoate in Treatment of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201546
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; DPI; Batefenterol; Fluticasone Furoate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — batefenterol; fluticasone furoate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Batefenterol + Fluticasone Furoate (Experimental): Subjects will self-administer batefenterol/fluticasone furoate 300/100 micrograms inhalation powder once daily for 42 days. Albuterol will be provided from screening to Day 42, to use as needed for symptom relief.
  Interventions: Drug: Batefenterol + Fluticasone Furoate; Drug: Albuterol
- Placebo (Placebo Comparator): Subjects will self-administer matching placebo inhalation powder once daily for 42 days. Albuterol will be provided from screening to Day 42, to use as needed for symptom relief.
  Interventions: Drug: Placebo; Drug: Albuterol

INTERVENTIONS:
Drug: Batefenterol + Fluticasone Furoate — Batefenterol and Fluticasone Furoate (FF) will be provided as a fixed-dose combination in a dry powder inhaler (DPI), for oral inhalation once every morning, for 42 days. The DPI will consist of 2 strips of 30 blisters each, containing 300 microgram (mcg) batefenterol per blister in one strip and 100 mcg FF per blister in another strip. Both drugs will be available in a micronized form, blended with lactose monohydrate.
  Arms: Batefenterol + Fluticasone Furoate
Drug: Placebo — Placebo will be provided in a DPI, for oral inhalation once every morning, for 42 days. The DPI will consist of 2 matching strips of 30 blisters each, with each blister containing lactose monohydrate and no active pharmaceutical ingredient.
  Arms: Placebo
Drug: Albuterol — Albuterol inhalation will be provided as an open-label rescue medication to use as needed, to relieve chronic obstructive pulmonary disease (COPD) symptoms.

SUMMARY:
Batefenterol inhalation powder is currently under development as a fixed-dose combination with fluticasone furoate (FF) for the treatment of Chronic Obstructive Pulmonary Disease (COPD).

The present study will administer batefenterol/FF (300/100 micrograms [mcg]) for the first time to subjects with COPD, to investigate the safety and tolerability of the combination compared with placebo, and to evaluate the pharmacokinetics and pharmacodynamics profiles of the individual components when administered in combination.

This is a Phase IIa, multicenter, randomized, placebo-controlled, double-blind, parallel group study. Subjects will be randomized (2:1) to one of the following double-blind treatment groups:

Batefenterol/FF 300/100 mcg inhalation powder once daily, or matching placebo inhalation powder once daily.

Subjects will self-administer the study treatments once daily (QD) in the morning for 42 days via a multi-dose dry powder inhaler (DPI) which contains two blister strips. Additionally, an inhaled short acting beta2-receptor agonist, albuterol will be provided from screening to the end of the treatment period for all subjects to use as needed to relieve COPD symptoms. At the end of the treatment period, subjects can resume conventional therapy.

The study will randomize approximately 60 subjects. The total duration of subject participation (from screening to follow-up) will be approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: Capable of giving signed informed consent, which includes compliance with pre-specified requirements and restrictions.
* Age and gender: Male and female subjects, 40 years of age or older at the time of signing the informed consent, are eligible to participate in the study.

Female subject: is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies:

1. Non-reproductive potential defined as:

   Pre-menopausal females with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; documented bilateral oophorectomy Postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
2. Reproductive potential and agrees to follow one of the options listed below 30 days prior to the first dose of study medication and until at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer after the last dose of study medication and completion of the follow-up visit. This list does not apply to females of reproductive potential with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis:

Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label Oral Contraceptive, either combined or progestogen alone Injectable progestogen Contraceptive vaginal ring Percutaneous contraceptive patches Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Chronic Obstructive Pulmonary Disease (COPD): An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* COPD Disease severity: A post-albuterol forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) ratio of =<0.70 and a post-albuterol FEV1 >=30 and =<80% of predicted normal values calculated using the European Respiratory Society Global Lung Function Initiative reference equations at Visit 1.
* Smoking history: Current or former cigarette smokers with a history of cigarette smoking of >= 10 pack-years at Visit 1. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.

Number of pack years = (number of cigarettes per day / 20) x number of years smoked (for example, 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years both equal 10 pack-years).

Note: Pipe and cigar use cannot be used to calculate pack-year history.

Exclusion Criteria:

* Asthma: A current diagnosis of asthma (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. Other excluded conditions include and not limited to clinically significant bronchiectasis, pulmonary hypertension unrelated to COPD, sarcoidosis, or interstitial lung disease. Or a subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Poorly controlled COPD: defined as the occurrence of 'acute worsening of COPD that is managed with corticosteroid and/or antibiotics or that requires treatment prescribed by a physician in the 6 weeks prior to Screening (Visit 1)', or 'subjects who are hospitalized due to acute worsening of COPD within 12 weeks of Visit 1'.
* History of COPD exacerbation: subject who have had more than one exacerbation (moderate or severe) within the 12 months prior to Visit 1.
* Pneumonia and lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Visit 1; or subjects hospitalized due to pneumonia within 12 weeks of Visit 1.
* Use of long-term oxygen therapy (LTOT): Oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (that is, =<12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (for example, albuterol) via nebulized therapy.
* Lung Resection: Lung volume reduction surgery within the 12 months prior to Visit 1.
* Clinically significant abnormal laboratory finding at Visit 1.
* Liver Disease: Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid polymerase chain reaction test is obtained.
* Abnormal and clinically significant findings from 12-lead electrocardiogram (ECG) performed at Visit 1. Site investigators will be provided with ECG over-read conducted by a centralized independent cardiologist, to assist in evaluation of subject eligibility. For this study, an abnormal and clinically significant ECG that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following:

Sinus bradycardia <45 beats per minute (bpm) (Note: Sinus bradycardia <45 bpm should be confirmed by two additional readings at least 5 minutes apart) Sinus tachycardia >=110 bpm (Note: Sinus tachycardia >=110 should be confirmed by two additional readings at least 5 minutes apart) Multifocal atrial tachycardia (wandering atrial pacemaker with rate >100 bpm) PR interval >240 milliseconds (msec) Evidence of Mobitz II second degree or third degree atrioventricular (AV) block Pathological Q waves (defined as wide [>0.04 seconds] and deep [>0.4 millivolt (mV) (4 millimeters [mm] with 10 mm/mV setting)] or >25% of the height of the corresponding R wave, providing the R wave was >0.5 mV [5 mm with 10 mm/mV setting], appearing in at least two contiguous leads (Note: prior evidence [that is, ECG obtained at least 12 months prior) of pathological Q waves that are unchanged are not exclusionary; and the investigator will determine if the subject is precluded from entering the study) Evidence of ventricular ectopic couplets, bigeminy, trigeminy or multifocal premature ventricular complexes.

For subjects without complete right bundle branch block: QT interval corrected by Fridericia's method (QTc[F]) >=450 msec or an ECG that is unsuitable for QT measurements (for example, poor defined termination of the T wave) For subjects with complete right bundle branch block: QTc(F) >=480msec or an ECG that is unsuitable for QT measurements (for example, poor defined termination of the T wave) (Note: All potentially exclusionary QT measurements should be confirmed by two additional readings at least 5 minutes apart) ST-T wave abnormalities (excluding non-specific ST-T wave abnormalities) (Note: prior evidence (that is, ECG obtained at least 12 months prior) of ST-T waves that are unchanged are not exclusionary and the investigator will determine if the subject is precluded from entering the study) Clinically significant conduction abnormalities (for example, Wolff-Parkinson-White syndrome or bifascicular block defined as complete left bundle branch block or complete right bundle branch block with concomitant left fascicular block) Clinically significant arrhythmias (for example, atrial fibrillation with rapid ventricular response, ventricular tachycardia)

* Medication Prior to Spirometry: Unable to withhold albuterol for the 4 hour period required prior to spirometry testing at each study visit.
* Excluded Medications: Use of the following medications are not permitted within the defined time intervals prior to Visit 1 and throughout the study:

Depot corticosteroids: 12 weeks Systemic, oral or parenteral corticosteroids: 6 weeks Antibiotics (for lower respiratory tract infection): 6 weeks 'Cytochrome P450 3A4' strong inhibitors and 'P-glycoprotein' inhibitor: 4 weeks Long acting beta-agonist (LABA)/inhaled corticosteroid (ICS) combination products : 4 weeks ICS : 4 weeks Phosphodiesterase 4 (PDE4) inhibitors (roflumilast): 1 week LABA/ Long-acting muscarinic antagonist (LAMA) combination (for example, vilanterol/umeclidinium bromide): 1 week Once-daily beta2-agonist (for example, Olodaterol and Indacaterol): 1 week LAMA (tiotropium, aclidinium, glycopyrronium, umeclidinium): 1 week Theophylline preparations: 48 hours Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton): 48 hours Oral beta2-agonists Long-acting: 48 hours Short-acting: 12 hours Inhaled LABA (for example, Salmeterol, formoterol): 48 hours Inhaled sodium cromoglycate or nedocromil sodium: 24 hours Inhaled short acting beta2-agonists: 4 hours Inhaled short-acting anticholinergics: 4 hours Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products: 4 hours Use of study provided albuterol is permitted during the study, except in the 4-hour period prior to spirometry testing

* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta-2-agonist, sympathomimetic, corticosteroid (intranasal, inhaled or systemic) lactose/milk protein, or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction, that, in the opinion of the study physician contraindicates study participation or use of an inhaled LAMA, LABA or ICS
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Affiliation with Investigator Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a diary.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2016-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (10):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Grove City, Ohio
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, McKinney, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20383

REFERENCES:
- [Background] Crim C, Gotfried M, Spangenthal S, Watkins M, Emmett A, Crawford C, Baidoo C, Castro-Santamaria R. A randomized, controlled, repeat-dose study of batefenterol/fluticasone furoate compared with placebo in the treatment of COPD. BMC Pulm Med. 2020 May 4;20(1):119. doi: 10.1186/s12890-020-1153-7. PMID 32366249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 1-week run-in period, 6-week (42-day) treatment period and 1-week follow-up period. Eligible participants (par.) were randomized (2:1) to either batefenterol (BAT)/fluticasone furoate (FF) 300/100 micrograms (µg) or a placebo in double blinded treatment.
Pre-assignment Details: A total of 62 participants withn an established clinical history of chronic obstructive pulmonary disease (COPD) were randomized and received at least one dose of study drug (forming the Intent-to-Treat Population), out of which 7 participants were withdrawn from the study.
Groups:
- Placebo: Participants received oral inhalation of placebo via a dry powder inhaler once daily in the morning for 6 weeks. Participants also received albuterol as a rescue medication throughout the study as needed, while receiving investigational product.
- BAT/FF 300/100 µg: Participants received oral inhalation of BAT/FF 300/100 µg via a dry powder inhaler once daily in the morning for 6 weeks. Participants also received albuterol as a rescue medication throughout the study as needed,while receiving investigational product.
Period: Overall Study
Arm/Group | Placebo | BAT/FF 300/100 µg
Started | 20 | 42
Completed | 20 | 35
Not Completed | 0 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other: Reached defined stopping criteria | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other: Fail to Meet Visit | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- BAT/FF 300/100 µg: Participants received oral inhalation of BAT/FF 300/100 µg via a dry powder inhaler once daily in the morning for 6 weeks. Participants also received albuterol as a rescue medication throughout the study as needed, while receiving investigational product.
- Total: Total of all reporting groups
Arm/Group | Placebo | BAT/FF 300/100 µg | Total
Number analyzed (Participants) | 20 | 42 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (8.86) | 63.0 (7.88) | 62.5 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 24 | 36
  Male | 8 | 18 | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 4 | 7
  American Indian or Alaskan Native | 1 | 0 | 1
  White - Arabic/North African Heritage | 0 | 2 | 2
  White - White/Caucasian/European Heritage | 16 | 36 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 0 to 4 Hours Post-dose Weighted Mean Heart Rate at Day 42, Derived From Electrocardiograms (ECGs)
Description: ECG measurements were taken in supine position after obtaining vital signs. Weighted mean was derived by calculating the area under the curve (AUC), and then dividing by the relevant time interval. Baseline was the pre-dose measurement on Day 1. Change from Baseline in 0 to 4 hours post-dose weighted mean heart rate was measured on Days 1, 28 and 42 and was analyzed using a mixed models repeated measures (MMRM) model. Intent-To-Treat (ITT) Population: all randomized participants who received at least one dose of study medication.
Time Frame: Baseline and Day 42
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Beats per minute (bpm)
Arm/Group | Placebo | BAT/FF 300/100 µg
Number analyzed (Participants) | 20 | 42
Beats per minute (bpm) | 0.688 (1.5238) | -1.557 (1.1374)
Statistical Analysis 1: Comparison: Placebo vs BAT/FF 300/100 µg; Test type: Non-Inferiority or Equivalence — p-values were not presented as non-inferiority was assessed by confidence interval (CI); Mean Difference (Final Values) = -2.245, 95% CI 2-sided [-6.153 to 1.663] — Treatment difference is calculated as active minus placebo and the non-inferiority bound was 10 bpm for Day 42

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected from start of the study until the follow-up contact (Visit 7 [Visit 6/EW +7 days]). Non-serious AEs were collected from the start of study treatment (Visit 2) until the follow-up contact (Visit 7)
Description: SAEs and non-serious AEs were reported for the ITT Population, comprised of all participants randomized to treatment and who received at least one dose of study medication. On-treatment AEs and SAEs were defined as those with onset between treatment start date and treatment stop date +1.
Arm/Group | Placebo | BAT/FF 300/100 µg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/42
Other Adverse Events (participants affected / at risk) | 7/20 | 8/42
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | BAT/FF 300/100 µg (N=42)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.